CLINICAL TRIAL: NCT06348745
Title: Trans Thoracic Ultrasound to Assess Diaphragmatic Function in Stable COPD Versus Bronchial Asthma.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Amer, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: diaphragmatic ultrasound
Record Dates: First submitted 2024-02-28; First posted 2024-04-05 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Diaphragm
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chronic obstructive pulmonary disease (COPD) (Experimental): ultrasound to COPD patients to asses' diaphragmatic function.
  Interventions: Device: ultrasound
- bronchial asthma (Experimental): ultrasound to bronchial asthma patients to asses' diaphragmatic function.
  Interventions: Device: ultrasound

INTERVENTIONS:
Device: ultrasound — 5. Transthoracic ultrasound for both right and left diaphragm during inspiration and expiration.

SUMMARY:
* Assessment of diaphragmatic function (excursion, thickness variation, thickness ratio) in COPD and bronchial asthma patients.
* Assessment of presence of correlation between diaphragmatic dysfunction and pulmonary function.
* Assessment of possible association between diaphragmatic dysfunction and presence of reversibility in pulmonary function post bronchodilator.

DETAILED DESCRIPTION:
* Assessment of diaphragmatic function (excursion, thickness variation, thickness ratio) in COPD and bronchial asthma patients.
* Assessment of presence of correlation between diaphragmatic dysfunction and pulmonary function (FEV1/FVC).
* Assessment of possible association between diaphragmatic dysfunction and presence of reversibility in pulmonary function post bronchodilator (short acting B2 agonist)

ELIGIBILITY:
Inclusion Criteria:

Stable patients (not in exacerbation).

Exclusion Criteria:

* Patients with comorbidities as cardiac, renal or hepatic diseases.
* Patients who have combined COPD and bronchial asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
diaphragmatic function | 2 years
  Compare diaphragmatic function using ultrasound device by measuring diaphragmatic thickness in both stable COPD and bronchial asthma patients.

SECONDARY OUTCOMES:
pulmonary function . | 2 years
  assess the degree of effect of diaphragmatic dysfunction on pulmonary function measured by spirometry FEV1/FVC (forced expiratory volume1/ forced Vidal capacity )

IPD SHARING:
Plan to Share IPD: No